CLINICAL TRIAL: NCT02606045
Title: Prospective, Randomized, Crossover Trial Comparing Recombinant Von Willebrand Factor (rVWF) vs. Tranexamic Acid (TA) to Minimize Menorrhagia in Women With Von Willebrand Disease: The VWD Minimize Study
Brief Title: Minimize Menorrhagia in Women With Von Willebrand Disease
Acronym: VWDMin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study stopped early due to slow recruitment.
Sponsor: Margaret Ragni (Other)
Collaborators: University of North Carolina (Other); Duke University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Margaret Ragni, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030221; U01HL133815 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-17 (Estimated); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Von Willebrand Diseases
Keywords: menorrhagia; VWD
MeSH Terms: conditions — von Willebrand Diseases; Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Subjects randomized to Group I will receive Arm A recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm B, tranexamic acid 650 mg 2 tablets orally (po) three times daily on days 1-5 of each of two menstrual cycles, Cycles 3 and 4.
  Interventions: Drug: recombinant von Willebrand factor; Drug: tranexamic acid
- Group II (Active Comparator): Group II will receive Arm B, tranexamic acid 650 mg 2 tablets orally (po) three times daily on days 1-5, for each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm A, recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 on each of two menstrual cycles, Cycles 3 and 4.
  Interventions: Drug: recombinant von Willebrand factor; Drug: tranexamic acid

INTERVENTIONS:
Drug: recombinant von Willebrand factor — Group I will receive Arm A recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm B, TA 650 mg 2 tablets orally (po) three times daily on days 1-5 of each of two menstrual cycles, Cycles 3 and 4.
  Group II will receive Arm B, TA 650 mg 2 tablets orally (po) three times daily on days 1-5, for each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm A, rVWF 40 IU/kg intravenously (IV) infusion on day 1 on each of two menstrual cycles, Cycles 3 and 4.
  Other Names: vonicog alfa; Vonvendi
Drug: tranexamic acid — Group I will receive Arm A recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm B, TA 650 mg 2 tablets orally (po) three times daily on days 1-5 of each of two menstrual cycles, Cycles 3 and 4.
  Group II will receive Arm B, TA 650 mg 2 tablets orally (po) three times daily on days 1-5, for each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm A, rVWF 40 IU/kg intravenously (IV) infusion on day 1 on each of two menstrual cycles, Cycles 3 and 4.
  Other Names: Lysteda®

SUMMARY:
This is an outpatient, 24-week Phase III prospective, randomized, crossover trial comparing recombinant von Willebrand factor (rVWF) and tranexamic acid (TA, Lysteda®) to minimize menorrhagia in women with von Willebrand disease (VWD). The purpose of this Phase III multicenter prospective, randomized, crossover arm trial is to compare recombinant von Willebrand factor (rVWF) to tranexamic acid (TA) in reducing the severity of menorrhagia in women with von Willebrand disease.

DETAILED DESCRIPTION:
In this study, women age 13-45 years with mild to moderate VWD and menorrhagia will be enrolled at their hemophilia treatment centers (HTCs) and provide information on menstrual bleeding from their two past monthly cycles to establish baseline bleeding frequency. Only women with regular menses, defined as menses every 21-35 days will be enrolled. A total of 60 subjects will be recruited and enrolled at approximately 25 HTC sites. Following enrollment, subjects will be randomized to Group I or Group II for the first five days of the next four consecutive menstrual cycles. Those randomized to Group I will be treated with Arm A for menstrual bleeding in cycles 1 and 2, followed by Arm B for menstrual bleeding in cycles 3 and 4. Those randomized to Group II will be treated with Arm B for menstrual bleeding in cycles 1 and 2, followed by Arm A for menstrual bleeding in cycles 3 and 4.

Subjects randomized to Group I will receive Arm A rVWF 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm B, TA 650 mg 2 tablets orally (po) three times daily on days 1-5 of each of two menstrual cycles, Cycles 3 and 4. Subjects randomized to Group II will receive Arm B, TA 650 mg 2 tablets orally (po) three times daily on days 1-5, for each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm A, rVWF 40 IU/kg intravenously (IV) infusion on day 1 on each of two menstrual cycles, Cycles 3 and 4. This regimen may be given at the HTC clinic or at home by visiting nurse. Baseline laboratory studies will be drawn at screening, including Blood Counts: hemoglobin, white count, differential, platelets; Iron Tests: iron, total iron binding capacity (TIBC), ferritin; Thyroid Test: thyroid stimulating hormone (TSH); and Von Willebrand Tests (VWF and related tests). Before initiating treatment, subjects will be trained by the HTC nurse on 1) reading urine pregnancy tests and 2) completion of the pictorial blood assessment chart (PBAC), cycle severity score (CSR), and cycle length (CL); and 3) completion of patient diary. Following randomization, subjects will administer home pregnancy tests prior to the first of each 5-day dosing cycle. On each of the four dosing cycles, Cycles 1-4, the PBAC, CSR, and CL will be recorded daily. After completion of study drug on cycle 2, the Crossover Study Visit will occur, during which subjects will be given a new supply of study drug for the study arm to which they will crossed over; subject diaries will be returned and coagulation studies and quality of life questionnaires performed. At 10-14 days after completion of study drug in Cycle 4, the End Study Visit will occur, during which subject diaries will be returned and quality of life questionnaires performed. All study visits will be within +/- 2 days of the scheduled visit. Study visits will be every 2 months, at the end of cycle 2 (cross-over) and at the end of cycle 4 (end of study) during which treatment diaries will be reviewed for bleeding frequency, side effects, and medications. Menstrual bleeding by PBAC, cycle severity, cycle duration, and health-related quality-of-life (HRQoL) questionnaires, including Rand Short Form 36-Question Health Survey (SF-36), Ruta Menorrhagia Severity Scale, Center for Disease Control Health-Related Quality of Life-14 Question Form (CDC-HRQoL14), and Center for Epidemiologic Studies Depression Scale (CES-D) will be assessed at baseline and after cycle 2 and after cycle 4. The study is innovative in the 1) evaluation of recombinant VWF, a new high purity recombinant VWF protein, to reduce menorrhagia, as compared with the current non-hormonal standard, tranexamic acid (TA); 2) investigation of the relationship of VWF to menstrual bleeding by PBAC score, by assessing VWD parameters: VWF ristocetin co-factor (VWF:RCo), VWF antigen (VWF:Ag), FVIII:C, VWF multimers, including high molecular weight multimers (HMW) by electrophoresis, and VWF genotype; 3) use of a "home treatment injection" for VWD; 4) comparison of two quality of life measures to assess treatment response on each study arm, one specific for bleeding disorders and one specific for menstrual disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females 13-45 years of age.
2. Mild or moderate von Willebrand disease (VWF:RCo <0.50 IU/ml, normal multimers, past bleeding)
3. Menorrhagia defined as PBAC >100 in at least one of the last two menstrual cycles.
4. Regular menses, at least every 21-35 days.
5. Willingness to have blood drawn
6. No prior history of an allergic reaction or anaphylaxis to rVWF or TA.
7. Willingness to avoid aspirin (ASA) and nonsteroidal anti-inflammatory agents (NSAIDS) during the study.
8. Willingness to comply with randomization to rVWF or TA study arms.
9. Willingness to keep a personal diary of menorrhagia bleeding frequency duration and severity by pictorial blood assessment chart, and any drugs or hemostatic agents taken.
10. Willingness to make 4 visits and undergo blood sampling for coagulation studies, and accept randomization of two therapies for each of four consecutive menstrual cycles, including an end-of-study visit.
11. Willingness to use "double-barrier" method of contraception during the study.

Exclusion Criteria:

1. Any bleeding disorder other than von Willebrand disease; or past thrombotic disease
2. Pregnant or lactating, or use of hormones (other than progesterone-only), or combined oral contraceptives, and contraceptive implants in past 3 months.
3. Platelet count < 100,000/ul.
4. Use of immunomodulatory or experimental drugs.
5. Surgery within the past 8 weeks.
6. Concomitant use of antiplatelet drugs, anticoagulants, dextran, aspirin or NSAIDs.
7. Treatment with DDAVP, cryoprecipitate, whole blood, plasma and plasma derivatives containing VWF within 5 days of study.
8. Inability to comply with study requirements.
9. Hypothyroidism as defined by elevated TSH.
10. Iron deficiency as defined by low serum ferritin, unless iron replacement has been initiated.
11. History of renal disease

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (19):
- United States (19):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Center for Inherited Blood Disorders (CIBD), Orange, California
  - University of California San Francisco, San Francisco, California
  - Emory University Afflac Blood Disorders Center, Atlanta, Georgia
  - Henry Ford Hospital Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Cure4thekids Foundation, Las Vegas, Nevada
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - State University of New York Upstate Medical Center, Syracuse, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh and Hemophilia Center Western PA, Pittsburgh, Pennsylvania
  - Vanderbilty University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Bloodworks Northwest, Seattle, Washington
  - Versiti Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The IPD to be shared include individual bleeding data (PBAC), cycle severity score (CSR), cycle length (CL), quality of life by four scales (SF-36, Ruta, CDC-HRQoL-14, CES-D), satisfaction survey, VWF assays, VWF genotype.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of trial completion.
Access Criteria: Qualified investigators will have access to data and bio specimens, consistent with data sharing policies and applicable laws, and upon receipt of a Research Materials Distribution Agreement, data will be transferred by secure transfers through the BioLINCC website.

REFERENCES:
- [Background] Ragni MV, Machin N, Malec LM, James AH, Kessler CM, Konkle BA, Kouides PA, Neff AT, Philipp CS, Brambilla DJ. Von Willebrand factor for menorrhagia: a survey and literature review. Haemophilia. 2016 May;22(3):397-402. doi: 10.1111/hae.12898. Epub 2016 Feb 4. PMID 26843404
- [Derived] Ragni MV, Rothenberger SD, Feldman R, Nance D, Leavitt AD, Malec L, Kulkarni R, Sidonio R Jr, Kraut E, Lasky J, Pruthi R, Angelini D, Philipp C, Hwang N, Wheeler AP, Seaman C, Machin N, Xavier F, Meyer M, Bellissimo D, Humphreys G, Smith KJ, Merricks EP, Nichols TC, Ivanco D, Vehec D, Koerbel G, Althouse AD. Recombinant von Willebrand factor and tranexamic acid for heavy menstrual bleeding in patients with mild and moderate von Willebrand disease in the USA (VWDMin): a phase 3, open-label, randomised, crossover trial. Lancet Haematol. 2023 Aug;10(8):e612-e623. doi: 10.1016/S2352-3026(23)00119-9. Epub 2023 Jun 26. PMID 37385272

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Von Willebrand Factor, Then Tranexamic Acid: Group I will receive Arm A recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm B, tranexamic acid 650 mg 2 tablets orally (po) three times daily on days 1-5 of each of two menstrual cycles, Cycles 3 and 4.
- Tranexamic Acid Then Recombinant Von Willebrand Factor: Group II will receive Arm B, tranexamic acid 650 mg 2 tablets orally (po) three times daily on days 1-5, for each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm A, recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 on each of two menstrual cycles, Cycles 3 and 4.
Period: Overall Study
Arm/Group | Recombinant Von Willebrand Factor, Then Tranexamic Acid | Tranexamic Acid Then Recombinant Von Willebrand Factor
Started | 18 | 21
Completed | 17 | 19
Not Completed | 1 | 2
Not completed — Study closed before treament could begin | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group I: Group I will receive Arm A recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, Cycles 1 and 2. They will then be crossed over to Arm B, tranexamic acid 650 mg 2 tablets orally (po) three times daily on days 1-5 of each of two menstrual cycles, Cycles 3 and 4.
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 4 | 4
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (6.3) | 26.7 (10.3) | 29.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36
Menstrual Bleeding Severity [Mean (Standard Deviation); unit: score on a scale] — As measured by Pictorial Blood Assessment Chart (PBAC), 0- no theoretical limit, higher score means greater severity
  score on a scale | 597 (389) | 483 (270) | 537 (331)

OUTCOME MEASURES:

1. Primary Outcome: Menstrual Bleeding Severity
Description: As measured by Pictorial Blood Assessment Chart (PBAC), 0- no theoretical limit, higher score means greater severity
Time Frame: 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tranexamic Acid: Participants who received tranexamic acid 650 mg 2 tablets orally (po) three times daily on days 1-5, for each of two menstrual cycles, in either first 2 cycle weeks of the study or the last 2 cycle weeks of the study
- Recombinant Von Willebrand Factor: Participants who received recombinant von Willebrand factor 40 IU/kg intravenously (IV) infusion on day 1 of each of two menstrual cycles, in either first 2 cycle weeks of the study or the last 2 cycle weeks of the study
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
score on a scale | 225 (207) | 272 (223)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Test type: Superiority; p = 0.039, Mixed Models Analysis; Mean Difference (Final Values) = 46, 95% CI 2-sided [2 to 90]

2. Secondary Outcome: Cycle Duration
Description: Menorrhagia cycle length by days of bleeding (score 0 - theoretically any length)
Time Frame: 4 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
days | 7.1 (4.5) | 7.0 (3.9)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Test type: Superiority; p = 0.998, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.7]

3. Secondary Outcome: Ruta Menorrhagia Severity Scale
Description: Unit measure derived from quality of life questions reported as a single score, Minimum 0 to 100 maximum, with a higher score indicating worse outcome
Time Frame: 4 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
units on a scale | 32.4 (13.5) | 34.8 (13.0)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Test type: Superiority; p = 0.168, Mixed Models Analysis; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-1.0 to 5.8]

4. Secondary Outcome: Center for Epidemiology Studies Depression Scale (CES-D)
Description: Reported by questions on depression, Minimum 0 to 60 Maximum, with higher scores indicating greater depression.
Time Frame: 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
score on a scale | 13.5 (10.6) | 11.0 (10.2)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Test type: Superiority; p = 0.055, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.9 to 0.1]

5. Secondary Outcome: Rand Short Form 36-Question Health Survey (SF-36)
Description: SF-36 reported by answer to questions, Minimum 0 to Maximum 100 for each of 8 domains (1-physical functioning, 2-role limitations due to physical health, 3-role limitations due to emotional problems, 4-energy and fatigue, 5-emotional wellbeing, 6-social functioning, 7-pain, and 8-general health), with higher scores for each domain meaning greater severity of physical and mental health.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
units on a scale
  Physical functioning | 84.4 (19.6) | 83.6 (20.0)
  Role limitations of physical health | 70.1 (39.1) | 67.4 (37.7)
  Role limitations of emotional health | 63.9 (41.7) | 68.5 (39.0)
  Energy/fatigue | 50.3 (20.6) | 47.9 (22.8)
  Emotional well-being | 69.2 (17.7) | 72.9 (20.0)
  Social functioning | 76.4 (21.9) | 80.9 (20.2)
  Pain | 71.2 (23.5) | 68.8 (34.2)
  General health | 58.8 (19.9) | 59.3 (21.2)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Test type: Superiority; p = 0.681, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-4.8 to 3.2]
Statistical Analysis 2: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Role limitations of physical health; Test type: Superiority; p = 0.633, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-12.4 to 7.6]
Statistical Analysis 3: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Role limitations of emotional health; Test type: Superiority; p = 0.362, Mixed Models Analysis; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-5.7 to 15.3]
Statistical Analysis 4: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Energy/fatigue; Test type: Superiority; p = 0.375, Mixed Models Analysis; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-7.4 to 2.8]
Statistical Analysis 5: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Emotional well-being; Test type: Superiority; p = 0.068, Mixed Models Analysis; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-0.3 to 7.4]
Statistical Analysis 6: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Social functioning; Test type: Superiority; p = 0.189, Mixed Models Analysis; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [-2.3 to 11.3]
Statistical Analysis 7: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Pain; Test type: Superiority; p = 0.489, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-9.2 to 4.5]
Statistical Analysis 8: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; General Health; Test type: Superiority; p = 0.786, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-3.2 to 4.3]

6. Secondary Outcome: Center for Disease Control Health-Related Quality of Life 14 Questions (CDC-HRQoL-14)
Description: Reported by answer to questions, over the past two weeks with minimum 0 to maximum 14, with higher scores indicating greater severity of physical and mental health.
Time Frame: 4 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
units on a scale
  Physically Unhealthy Days | 3.1 (4.0) | 1.9 (3.2)
  Mentally Unhealthy Days | 4.7 (5.1) | 5.7 (7.0)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Physically Unhealthy Days; Test type: Superiority; p = 0.098, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.3 to 0.2]
Statistical Analysis 2: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Mentally Unhealthy Days; Test type: Superiority; p = 0.557, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.6 to 3.0]

7. Secondary Outcome: Cycle Severity
Description: Menorrhagia cycle severity by Likert scale, with minimum 0 to maximum 3, with higher score indicating worse severity.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
Number analyzed (Participants) | 36 | 36
units on a scale | 0.96 (0.879) | 1.07 (0.738)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Recombinant Von Willebrand Factor; Cycle Severity Rating; Test type: Superiority; p = 0.266, Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.8 to 2.7]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over collected a 24 week period
Description: Includes all participants who received study intervention
Arm/Group | Tranexamic Acid | Recombinant Von Willebrand Factor
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 4/36 | 4/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=36) | Recombinant Von Willebrand Factor (N=36)
Mucosal Bleeding (Blood and lymphatic system disorders) | 2 (4) | 0 (0) — mucosal bleeding in the oropharyngeal, gastrointestinal, and genitourinary tracts
Other Bleeding (Blood and lymphatic system disorders) | 3 (4) | 2 (2) — vaginal bleeding
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Injury/ Trauma Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Brusing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT02606045/Prot_SAP_003.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT02606045/ICF_002.pdf